CLINICAL TRIAL: NCT03364452
Title: The Validation of Various Dietary Assessment Methodologies
Status: Completed | Type: Observational
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Valisa Hedrick, Assistant Professor, Virginia Polytechnic Institute and State University
Other Study IDs: Diet Assessment Methods
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Diet Habit
Keywords: Dietary Assessment Methodology; beverages; non-nutritive sweeteners
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is see how well two dietary intake questionnaires, blood values, and urine samples can estimate what participants are eating and drinking. Specifically, the investigators are looking at the validity of a new artificial sweetener food frequency questionnaire and a urinary biomarker for artificial sweetener consumption. Additionally, the investigators are examining the ability of a rapid beverage intake questionnaire (BEVQ-15) to determine Healthy Beverage Index scores.

DETAILED DESCRIPTION:
The role of beverages in overall dietary patterns and health is controversial but remains an important key target for clinical interventions and public policy. Additionally, non-nutritive sweetener intake is controversial. It is difficult to measure intake; therefore, it is difficult to determine associations to health outcomes. For this study, the investigators plan to study 125 adult participants during 3 visits over 2 weeks. The purpose of this study is two-fold: 1) to assess the utility of two food frequency questionnaires (the Healthy Beverage Index and the Non-Nutritive Sweetener questionnaire) and 2) to assess the capabilities of a non-nutritive sweetener biomarker.

The first goal of this study is to assess the validity of the Healthy Beverage Index (HBI) via the BEVQ-15 questionnaire compared to the HBI via dietary recalls. Additionally, the correlations of HBI scores to dietary intake biomarkers will be assessed (urinary specific gravity) and associations between HBI scores with weight status and related cardio-metabolic health variables will be determined (weight, blood pressure, waist circumference, blood lipids, and glucose). The investigators will assess potential confounds to the HBI (health literacy, socio-economic status, demographics). The second goal is to assess the correlations between the non-nutritive sweetener food frequency questionnaire and the 24-hour dietary recalls.

The investigators predict that 1) HBI scores will not vary significantly between BEVQ-15 and dietary recall assessment methods, 2) HBI scores will be significantly correlated to the dietary biomarker (negative association between urinary specific gravity and total fluid intake), 3) there will be statistically significant relationships between HBI scores and health indicators, and 4) non-nutritive sweetener consumption reported in the non-nutritive sweetener questionnaire and the 24-hour dietary recalls will be significantly correlated.

ELIGIBILITY:
Inclusion Criteria:

* The subject pool for this study includes adults. Participants must be 18 years of age or older and must speak English.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The aim of this project is to study dietary consumption patterns and identify a method to assess habitual non-nutritive sweetener consumption in the adult population (food frequency questionnaire and biomarker). Thus, our study aims to recruit a sample of participants that represents the general population.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
non-nutritive sweetener intake | 2 weeks
  agreement between non-nutritive sweetener intake from the food frequency questionnaire and dietary recalls and between the urinary biomarker and dietary recalls
Healthy Beverage Index Scores | 2 weeks
  Healthy Beverage Index scores are similar to Healthy Eating Scores and range from 0-100, with higher scores indicating greater agreement with beverage recommendations and guidelines. Agreement between total Healthy Beverage Index Scores from the BEVQ-15 (a beverage frequency questionnaire) and Healthy Beverage Index Scores from dietary recalls will be compared.

SECONDARY OUTCOMES:
Metabolic syndrome and non-nutritive sweetener intake | 2 weeks
  Association between metabolic syndrome incidence and non-nutritive sweetener intake

CONTACTS AND LOCATIONS:
Overall Officials: Valisa E Hedrick, PhD, RDN, Principal Investigator — Virginia Polytechnic Institute and State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hess EL, Myers EA, Swithers SE, Hedrick VE. Associations Between Nonnutritive Sweetener Intake and Metabolic Syndrome in Adults. J Am Coll Nutr. 2018 Aug;37(6):487-493. doi: 10.1080/07315724.2018.1440658. Epub 2018 Mar 30. PMID 29601264